CLINICAL TRIAL: NCT02765568
Title: Investigating the Effects of Cardiac Rehabilitation eXercise Modalities on Physical and Mental Health Outcomes
Acronym: CRX-Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20160127-01H
Record Dates: First submitted 2016-04-29; First posted 2016-05-06 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention (PCI)
MeSH Terms: conditions — Coronary Artery Disease | interventions — High-Intensity Interval Training; Nordic Walking

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Moderate Intensity Continuous Exercise (Experimental): Moderate Intensity Continuous Exercise Training
  Interventions: Behavioral: Moderate Intensity Continuous Exercise Training
- Nordic Walking (Experimental): Nordic Walking
  Interventions: Behavioral: Nordic Walking
- High Intensity Interval Training (Experimental): High Intensity Interval Training
  Interventions: Behavioral: High Intensity Interval Training

INTERVENTIONS:
Behavioral: High Intensity Interval Training — Participants will complete supervised exercise sessions. Participants will attend on-site high-intensity interval training two times weekly for 12 weeks
  Other Names: HIIT
  Arms: High Intensity Interval Training
Behavioral: Moderate Intensity Continuous Exercise Training — Participants will complete supervised exercise sessions. Moderate-intensity continuous exercise training will follow cardiovascular rehabilitation guidelines. Participants will attend on-site moderate-intensity continuous exercise training two times weekly for 12 weeks.
  Other Names: MICE
  Arms: Moderate Intensity Continuous Exercise
Behavioral: Nordic Walking — Participants will complete supervised exercise sessions. Participants will attend on-site Nordic walking training two times weekly for 12 weeks
  Other Names: NW
  Arms: Nordic Walking

SUMMARY:
Coronary revascularization improves survival for patients with coronary artery disease. However,many patients are left with poor physical and mental health. Traditional cardiac rehabilitation involves moderate intensity continuous exercise (MICE). Alternatives to traditional cardiac rehabilitation programming may however provide superior understudied benefits to patients with poor physical and mental health. Nordic walking (NW) and high-intensity interval training (HIIT) are two examples of alternative programs for cardiac rehabilitation, which may provide superior physical and mental health benefits when compared to traditional MICE. The main purpose of this project is, therefore, to determine the short and long term physical and mental health benefits of alternative cardiac rehabilitation modalities, including NW and HIIT on exercise capacity, quality of life and depression after a 12-week program.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CAD who recently underwent PCI (within 2-10 weeks) PCI or coronary artery bypass grafting (within the last 18 weeks);
* Patient is referred to University of Ottawa Heart Institute cardiac rehabilitation program;
* Patient is able to walk independently
* Patient is willing to attend an onsite cardiac rehabilitation program twice weekly for 12 weeks;
* At least 40 years of age;
* Patient is willing and able to provide informed consent

Exclusion Criteria:

* Currently participating in routine exercise training (>2x/week) and/or using Nordic Walking poles;
* Active infection or inflammatory condition;
* Over 75 years of age;
* Persistent or permanent atrial fibrillation;
* Pregnant, lactating or planning to become pregnant during the trial period;
* Unstable angina or established diagnosis of chronic obstructive pulmonary disease, severe mitral or aortic stenosis, or hypertrophic obstructive cardiomyopathy;
* Unable to read and understand English or French;
* Unwilling or unable to return for follow-up visit at weeks 12 and 26;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in exercise capacity from baseline to 12 weeks and baseline to 26 weeks are measured by the six-minute walk test

SECONDARY OUTCOMES:
Functional Fitness | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in functional fitness from baseline to 12 weeks and baseline to 26 weeks are measured by the Senior Fitness Test
Aortic stiffness | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in aortic stiffness from baseline to 12 weeks and baseline to 26 weeks are measured by pulse wave velocity
Body Composition | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by the waist circumference.
Body Composition | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by bioelectrical impedance.
Body Composition | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in body composition from baseline to 12 weeks and baseline to 26 weeks are measured by body mass index.
Depression | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in depression from baseline to 12 weeks and baseline to 26 weeks are measured by the Beck Depression Inventory-II questionnaire
Quality of Life - SF36 | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in quality of life from baseline to 12 weeks and baseline to 26 weeks are measured by the Short Form-36.
Quality of Life - HeartQoL | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in quality of life from baseline to 12 weeks and baseline to 26 weeks are measured by the HeartQoL questionnaire
Exercise Adherence | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in exercise adherence from baseline to 12 weeks and baseline to 26 weeks are measured by the Actigraph accelerometer
Depression mechanisms | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in depression mechanisms from baseline to 12 weeks and baseline to 26 weeks are measured by plasma brain derived neurotrophic factor.
Depression mechanisms | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in depression mechanisms from baseline to 12 weeks and baseline to 26 weeks are measured by plasma irisin.
Depression mechanisms | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in depression mechanisms from baseline to 12 weeks and baseline to 26 weeks are measured by plasma kynurenine.
Lipid and glucose profile | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in lipid and glucose profile from baseline to 12 weeks and baseline to 26 weeks are measured by plasma total cholesterol.
Lipid and glucose profile | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in lipid and glucose profile from baseline to 12 weeks and baseline to 26 weeks are measured by plasma Low Density Lipoprotein
Lipid and glucose profile | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in lipid and glucose profile from baseline to 12 weeks and baseline to 26 weeks are measured by plasma High Density Lipoprotein.
Lipid and glucose profile | Baseline to 12 weeks and Baseline to 26 weeks
  Changes in lipid and glucose profile from baseline to 12 weeks and baseline to 26 weeks are measured by plasma Hemoglobin A1c

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Insititue, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marcal IR, Cotie LM, Ribeiro I, Reed JL. The Effects of Different Exercise Modalities and Intensities on Arterial Stiffness in Patients With Coronary Artery Disease. J Cardiopulm Rehabil Prev. 2023 Sep 1;43(5):384-385. doi: 10.1097/HCR.0000000000000799. Epub 2023 May 15. No abstract available. PMID 37184470
- [Derived] Garneau L, Terada T, Mistura M, Mulvihill EE, Reed JL, Aguer C. Exercise training reduces circulating cytokines in male patients with coronary artery disease and type 2 diabetes: A pilot study. Physiol Rep. 2023 Mar;11(5):e15634. doi: 10.14814/phy2.15634. PMID 36905198